CLINICAL TRIAL: NCT04775602
Title: Experimental Study to Evaluate the Impact of 18F-PSMA PET / CT in the Management of Patients with Prostate Cancer.
Brief Title: Experimental Study to Evaluate the Impact of 18 Fluoro-PSMA (18F-PSMA) PET / CT in the Management of Patients with Prostate Cancer.
Acronym: F-PSMA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRST185.07; 2019-002000-41 (EudraCT Number)
Record Dates: First submitted 2020-01-21; First posted 2021-03-01 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: 18F-PSMA; Prostate Cancer
Keywords: 18F-PSMA; PET/CT; Prostate Cancer; Diagnostic; Biochemical relapse; Negative standard imaging; Radically treated
MeSH Terms: conditions — Prostatic Neoplasms; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 18F-PSMA PET/CT (Experimental): Patients with evidence of biochemical recurrence of prostate cancer radically treated, with negative results to traditional diagnostic methods or doubtful imaging of 18F- Fluoro Methyl Choline (18F-FMC) PET/CT will perform a 18F-PSMA PET/CT as a tool for searching and location of recurrence.
  Interventions: Drug: 18F-PSMA

INTERVENTIONS:
Drug: 18F-PSMA — 18F-PSMA will be injected intravenously at a dosage of 200-250 megabecquerel (MBq) prior to perform Image acquisition (Topogram, CT, PET)

SUMMARY:
Single-center, prospective, open-label, not randomized, diagnostic phase II trial in the management of patients with prostate cancer.

DETAILED DESCRIPTION:
Single-center, prospective, open-label, not randomized, diagnostic phase II trial in the management of patients with prostate cancer. The aim of this study is to evaluate the additional diagnostic role of 18F- PSMA PET /CT (sensitivity) in patients with prostate cancer with biochemical relapse compared to other diagnostic methods routinely used. The primary objective is to evaluate the sensitivity of 18F-PSMA PET/CT defined as the ratio between the number of 18F-PSMA PET/CT positive patients and the number of prostate cancer patients with biochemical relapse and negative standard imaging.Patients enrolled in the study would benefit from a more accurate but above all earlier diagnosis of disease recurrence sites, thus being able to undergo targeted therapies, with a clear impact on the clinical management of the disease.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed prostate cancer
2. Male, aged >18 years on the day of signing and dating the informed consent form.
3. Previous radical treatment for prostate cancer (radiotherapy or surgery)
4. Negativity of all the other traditional morphological and functional imaging or doubtful imaging of 18F-FMC PET/CT
5. Patients with PSA progression defined as PSA ≥ 0.2 ng/mL and PSA rising defined as 2 subsequent values showing PSA increase at least 1 week apart.
6. Male participants whose partner is of child bearing potential must be willing to ensure that they or their partner use effective contraception during the study and for 3 months thereafter
7. Participant is willing and able to give informed consent for participation in the study.

Exclusion Criteria:

1. Hormonotherapy in the last 6 months
2. No radiotherapy in the last 6 months.
3. Participation in another clinical trial with any investigational agents within 30 days prior to prior informed consent date
4. History of allergic reactions attributed to compounds of similar chemical or biologic composition to Study Agent.
5. Medical or psychological conditions that would not permit the subject to sign the informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2020-07-31 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2024-07-11 (Actual)

PRIMARY OUTCOMES:
Diagnostic role of 18F- PSMA PET /CT (sensitivity) | Up to 30 months
  Sensitivity of 18F-PSMA PET/CT will be calculated as the ratio between the number of 18F- PSMA PET/CT positive patients and number of patients with radically treated prostate cancer with biochemical relapse and negativity of traditional morphological imaging.

SECONDARY OUTCOMES:
Sensitivity for different PSA values (ranges) | Up to 30 months
  Sensitivity of 18F-PSMA PET/CT will be stratified respect to different ranges of Prostate-Specific Antigen (PSA) values.
Sensitivity for different lesion sites | Up to 30 months
  Sensitivity of 18F-PSMA PET/CT will be stratified respect to different sites of lesion.
predictive role of 18F-PSMA PET/CT on disease status according to standard imaging and PSA evaluation. | Up to 30 months
  To evaluate the predictive role of 18F-PSMA PET/CT on disease status, for patients that will start an anticancer treatment. It will be performed the receiver operating characteristic (ROC) curves generated by plotting sensitivity versus 1-specificity The best cut-off value for distinguishing between positive and negative 18F- PSMA PET/CT findings will be determined using Youden's index.
evaluation of the concordance between 18F-PSMA PET/CT and other methods | Up to 30 months
  To evaluate the concordance between 18F-PSMA PET/CT and PET/CT or the others standard methods, for patients without any treatment, it will be performed by Cohen's kappa coefficient
18F-PSMA Safety: treated patients undergoing grade 1 to 4 adverse event | Up to 30 months
  Number and percentage of treated patients undergoing grade 1 to 4 adverse events will be tabulated according to CTCAE version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Federica Matteucci, MD, Principal Investigator — IRST IRCCS, Meldola (FC)
Locations (1):
- Irst Irccs, Meldola, FC, Italy

IPD SHARING:
Plan to Share IPD: Undecided